CLINICAL TRIAL: NCT02167841
Title: Comparison of Efficiency Between Practicing of Knee Chest Position and External Cephalic Version in Cases of Breech Presentation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0265-13-MMC
Record Dates: First submitted 2014-06-11; First posted 2014-06-19 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Breech Presentation
Keywords: Breech presentation,; External cephalic version,; Maternal posture,; Pregnancy,; Caesarean section.
MeSH Terms: conditions — Breech Presentation | interventions — Knee-Chest Position

ARMS (2):
- Knee-Chest position (Experimental): In this arm, the women will perform daily the Knee-Chest position between weeks 32-37. In week 37 the investigators will check via ultra sound if there was a successful version (if not, the woman would go to External Cephalic Version)
  Interventions: Behavioral: Knee-Chest Position
- External Cephalic Version (No Intervention): In this group the women will perform External Cephalic Version without doing maternal Knee-Chest position before.

INTERVENTIONS:
Behavioral: Knee-Chest Position
  Arms: Knee-Chest position

SUMMARY:
Background: The incidence of breech presentation in pregnant women is 4%. The situation can be treated by two methods. The first is a version of the fetus from breech presentation to head presentation, which can be performed in several ways, such as, an action called EXTERNAL CEPHALIC VERSION as well as the Knee-Chest position by the pregnant mother and the second is a cesarean section. In this study we wish to investigate if the Knee-Chest position is as effective as the ECV action and as a result to decrease the need for ECV.

Hypotheses: According to our assumption, the Knee-Chest position can reduce the need for the ECV action.

Objectives: Investigate whether daily Knee-Chest position is as effective as ECV.

Methods: The investigators will conduct a "randomized clinical trial" study. Every pregnant woman in a breech presentation with a singleton between weeks 28-32 will be randomly assigned into one of two groups. In the first group the women will perform daily the Knee-Chest position between weeks 32-37. In week 37 the investigators will check via ultra sound if there was a successful version (if not, the woman would go to ECV) in the second group we will perform ECV without doing maternal Knee-Chest position before. Every woman will fill a questionnaire which includes gynecological history and details regarding the degree of persistence and performance of the activity. At the end of this process the investigators will analyze the results and will come to the conclusions.

Significance: With ECV there are number of risks and complications such as fetal distress, placental abruption, rupture of membrane, amniotic fluid embolism or damage to the uterus. The frequency of these complications is 1%-2%. If it is discovered that the Knee-Chest position is effective as the ECV action, the investigators will recommend every patient to persist with this position and avoid the ECV action and the risks it entails.

ELIGIBILITY:
Inclusion Criteria:

Pregnant woman in a breech presentation with a singleton between weeks 28-32.

Exclusion Criteria:

* Antepartum Hemorrhage.
* Premature rupture of membranes.
* Placenta Previa.
* Oligohydramnios.
* Twin Pregnancy.
* Uterine malformation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
number of participants | up to 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Hospital, Kfar Saba, Israel